CLINICAL TRIAL: NCT00315016
Title: Eplerenone, ACE Inhibition and Albuminuria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRG 2005-316
Record Dates: First submitted 2006-04-14; First posted 2006-04-17 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Diabetic Nephropathy
Keywords: albuminuria; eplerenone; ACE inhibition; renal function; endothelial function
MeSH Terms: conditions — Diabetic Nephropathies; Albuminuria | interventions — Eplerenone; Fosinopril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): placebo (double dummy)
  Interventions: Drug: placebo
- 2 (Active Comparator): eplerenone
  Interventions: Drug: eplerenone
- 3 (Active Comparator): doubling of fosinopril dose
  Interventions: Drug: fosinopril

INTERVENTIONS:
Drug: eplerenone — active comparator
  Other Names: Eplerenone or INSPRA
  Arms: 2
Drug: fosinopril — doubling of fosinopril dose
  Other Names: fosinopril or Newace
  Arms: 3
Drug: placebo — placebo (double dummy)
  Other Names: no other name
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether eplerenone is more effective than doubling the dose of ACE inhibitor in reducing urinary protein (albumin) loss in diabetes mellitus

DETAILED DESCRIPTION:
In patients with proteinuric renal diseases renal function almost invariably deteriorates, independent from the original renal disease. It has been demonstrated that the rapidity of renal function deterioration is determined by blood pressure and proteinuria1. Treatment modalities that lower proteinuria in general tend to attenuate the deterioration of renal function. As such, ACE-inhibitors have been proven to be of particular value in the treatment of patients with proteinuria, since these drugs consistently lower proteinuria. More recently, similar antiproteinuric effects have been described for the angiotensin receptor blockers (ARBs). Theoretically, ACE inhibitors may have advantages over ARBs because they are supposed to increase bradykinin levels. Bradykinin has also been implicated in the development of nephropathy in mice. About its role in human diabetic nephropathy few if any data exist. The effect of ACE inhibition or ARBs is not complete, since addition of either drug to the other may further improve albuminuria. This may be explained by insufficient dosage of single drug therapy or because of an escape phenomenon. The latter has been amply described for ACE inhibitors. Especially with chronic ACE inhibition angiotensin II levels may be near normal. This may lead to persistent angiotensin II effects, among which aldosterone stimulation.

Even though most investigators have emphasized the role of the renin-angiotensin system in progressive renal injury, aldosterone has received little attention. However, its profibrotic effects make aldosterone a potentially important player in the field, even more so because the escape of aldosterone during treatment with ACE-inhibitors or ARBs. Moreover, in addition to these theoretical considerations, evidence is emerging that mineralocorticoid receptor blockade with spironolactone added to ACE-inhibitors or ARBs indeed has an additive, favourable effect on proteinuria. These findings warrant a search for the value of such agents in albuminuria and exploration of the mechanisms by which mineralocorticoid blockade may exert its beneficial effects.

Primary aim:

1. To study whether the combination of eplerenone and a standard dose of ACE-inhibition has an additive effect on albuminuria in patients with albuminuric nephropathy compared to ACE-I alone, or double dose of ACE-inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* documented diabetic renal disease with albuminuria >0.020 g/L, stable renal function (i.e. increase of serum creatinine <25% / 6 months), creatinine clearance > 40 ml/min/1.73 m2 , in spite of maximal ACE-inhibition (40 mg fosinopril/day)
* blood pressure < 140/90 mm Hg ( at baseline)
* serum potassium < 5.0 mmol/l (at baseline).

Exclusion Criteria:

* use of NSAID's or immunosuppressive drugs
* use of ARBs, intolerance for ACE inhibition.
* use of diuretics that increase potassium such as triamterene, spironolactone or eplerenone
* pregnancy
* rash or cough on one on the drugs
* severe heart disease or instable angina

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
proteinuria | 0, 4, 12, 24 and 30 weeks
blood pressure by home measurements | 0, 4, 12, 24 and 30 weeks

SECONDARY OUTCOMES:
serum potassium | 0, 3, days, 2, 4, 12, 24 and 30 weeks
haemoglobin | 0, 4, 12, 24 and 30 weeks
urinary excretion of CTGF, TGF-b, collagen IV | 0, 4, 12, 24 and 30 weeks
inulin and PAH clearance | 0, 24 and 30 weeks
Quality of Life | 0, 4, 12, 24 and 30 weeks
plasma aldosterone, renin | 0, 24 and 30 weeks
plasma angiotensins and bradykinins | 0, 24 and 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Deinum, MD, Principal Investigator — University Medical Center Nijmegen St Radboud, The Netherlands
Locations (2):
- Netherlands (2):
  - Jeroen Bosch Hospital, 's-Hertogenbosch, North Brabant
  - University Medical Center Nijmegen St Radboud, Nijmegen

REFERENCES:
- [Derived] Chung EY, Ruospo M, Natale P, Bolignano D, Navaneethan SD, Palmer SC, Strippoli GF. Aldosterone antagonists in addition to renin angiotensin system antagonists for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2020 Oct 27;10(10):CD007004. doi: 10.1002/14651858.CD007004.pub4. PMID 33107592